CLINICAL TRIAL: NCT00991432
Title: An Open Label, Non-randomized, Single-arm, Multi-center Study to Assess Localized Alveolar Ridge Augmentation Utilizing INFUSE® Bone Graft Concurrent With Space Maintenance Devices for Soft Tissue Management
Brief Title: Localized Alveolar Ridge Augmentation With Space Maintenance Devices
Acronym: Ridge Mesh
Status: Terminated | Type: Observational
Sponsor: Medtronic Spinal and Biologics (Industry)
Collaborators: Averion International Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: P09-04
Record Dates: First submitted 2009-10-06; First posted 2009-10-08 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2011-09

CONDITIONS: Alveolar Bone Loss
Keywords: Alveolar Ridge Augmentation; Dental Implantation, Endosseous; Osseointegration; Space Maintenance; Bone Morphogenetic Proteins
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- INFUSE® Bone Graft: all study participants will receive INFUSE® Bone Graft
  Interventions: Device: INFUSE® Bone Graft

INTERVENTIONS:
Device: INFUSE® Bone Graft — Patients will be treated with the commercially available INFUSE® Bone Graft material applied to an ACS concurrent with space maintenance devices for soft tissue management on Day 0 (Surgery). A follow-up visit will take place 2 weeks after implant of the INFUSE® Bone Graft material, or as regularly scheduled as per the standard of care (SOC) for the facility. Patients will return to the facility for final End of Study (EOS) assessments approximately 6 months after surgery. Between the follow-up visit and the EOS visit, patients will be seen as per the SOC schedule for the facility.

SUMMARY:
The purpose of this research study is to determine whether this study treatment can improve the bone structure of the upper front part of the jaw in patients who are scheduled for surgery to have a dental implant(s) placed into the upper front part of their mouths and need to have more bone in their jaws to support the implant, so that a dental implant can later be inserted.

DETAILED DESCRIPTION:
The INFUSE® Bone Graft is a device approved by the FDA to be used instead of using your own bone (from another site on your body) to replace missing bone in your jaw. INFUSE® Bone Graft is commercially available and is made up of 2 parts - recombinant human Bone Morphogenetic Protein-2 (rhBMP 2) placed on an absorbable collagen sponge (ACS). The rhBMP-2 is a genetically altered protein which recruits bone-forming cells to the surgical area and changes local cells to bone. ACS is made from Type I collagen from bovine (cattle) tendon. It helps to hold the rhBMP-2 in place and acts as a support for the growing bone. The sponge itself will reabsorb in time as the new bone forms.

The purpose of this research study is to determine whether this study treatment can improve the bone structure of the upper front part of the jaw so that a dental implant can later be inserted. This post-market study has been designed to further evaluate the effectiveness and safety of INFUSE® Bone Graft, along with space holding devices, in a 2-part procedure. Your dental implants will be placed at approximately 6 months after the INFUSE® Bone Graft implant.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent
2. ≥ 18 years
3. Scheduled for dental implant into anterior maxillary alveolar ridge
4. Negative urine pregnancy test for patients of child bearing potential and agreement not to become pregnant for at least 12 months after surgery
5. Able to comply with all study-related procedures, including exercising good oral hygiene
6. A prosthodontic treatment plan has been drafted.

Exclusion Criteria:

1. Known hypersensitivity to rhBMP-2, bovine Type I collagen or other components of the formulation
2. Known hypersensitivity to titanium
3. Operative site is in the area of a resected or extant tumor
4. Any active malignancy or current treatment for a malignancy
5. Active infection at operative site
6. History of prior exposure to rhBMP-2/ACS
7. Received and failed a previous alveolar ridge augmentation procedure
8. Pathology that would either compromise a bone grafting procedure, or interfere with obtaining quantitative measurements from postoperative computer tomography scans
9. Significant untreated periodontal disease (> Grade III), caries, or chronic inflammation of the oral cavity at operative site
10. Active use of any nicotine-containing products such as, but not limited to, smoking and chewing tobacco, nicotine patch, nicotine gum, etc.
11. Insulin-dependent diabetic, or has known glycated hemoglobin (HgbA1c) levels >6.5 %
12. History of malignancy within the past 5 years except for basal cell or squamous cell carcinoma of the skin
13. Patients who are lactating
14. History of metabolic bone disease, excluding idiopathic osteoporosis
15. History of autoimmune disease (e.g., documented multiple allergies, systemic lupus erythematosus, dermatomyositis, etc.) or immunosuppressive disease (e.g., human immunodeficiency virus or acquired immunodeficiency syndrome)
16. History of immune deficiency due to other treatments (e.g., radiation therapy, chemotherapy, steroid therapy)
17. History of adverse reaction to prior exposure to silicone or injectable collagen
18. Treatment with an investigational therapy within 1 month before the surgical procedure or plans to be treated with an investigational therapy during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients needing bone augmentation of the alveolar ridge
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Alveolar ridge bone formation sufficient to place endosseous implants | approximately 6 months post-surgery

SECONDARY OUTCOMES:
Evidence of successful INFUSE® Bone Graft placement, an increase in the alveolar ridge width and the safety of INFUSE® as assessed by CT scans. | approximately 6 months post-surgery

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Los Angeles, California
  - Greenwood Village, Colorado
  - Sarasota, Florida
  - Chicago, Illinois
  - Lafayette, Indiana
  - Denver, North Carolina
  - Portland, Oregon